CLINICAL TRIAL: NCT00276471
Title: Evaluation of the Tantalus System in Type 2 Diabetic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MetaCure Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC PT TAN2005-013
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Electrodes

INTERVENTIONS:
Device: Implantable pulse generator and electrodes

SUMMARY:
Metacure MC PT TAN2005-013 feasibility study is a prospective, multi-center, study to evaluate the safety and functionality of the TANTALUS System, in the treatment of obese T2DM patients, and to assess the effect of GCT ( Glycemic Control Treatment )on weight loss and glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* T2DM subjects inadequately controlled on a maximum of three oral agents
* Subjects with HbA1c between 7 and 9%
* Subjects with FBG between 120 and 200 mg/dL
* Subjects who are 21-60 years old
* Women with childbearing potential (i.e. not post-menopausal or surgically sterilized) must agree to use adequate birth control methods and must agree not to conceive for at least 20 weeks
* Subjects with Body Mass Index (BMI) between 30-38 (inclusive)
* Subjects with waist circumference >94 cm (males) and >80 cm (females)
* Subjects on stable medication program for at least three months with any oral medication program
* Subjects who are compliant, willing and able to participate in the follow-up visits for the study duration of approximately 26 weeks
* Alert, mentally competent, and able to understand and comply with the requirements of the clinical trial, and be personally motivated to abide by the requirements and restrictions of the clinical trial.
* Able to provide voluntary informed consent.

Exclusion Criteria:

* Subjects at high risk of general anesthesia or surgery
* Subjects with prior pancreatitis
* Subjects with chronic hepatitis
* Subjects with elevated serum creatinine
* Subjects with proliferative diabetic retinopathy
* Subjects with gastroparesis or intestinal pseudo-obstruction
* Subjects with motility disorders of the GI tract
* Subjects who are receiving medications known to affect gastric motility
* Subjects with a past or present psychiatric condition that may impair his or her ability to comply with the study procedures
* Subjects who are pregnant (proven by positive hCG), or lactating
* Subjects who have had prior bariatric surgery
* Subjects with a history of peptic ulcer disease
* Subjects who have used another investigational device or agent in the 30 days prior to implant or are participating in any other clinical study
* Subjects with any new medical problem diagnosed or the worsening of an existing medical problem during the baseline evaluation period
* Subjects with a life-threatening co-morbidity or life expectancy of less than one year
* Subjects with myocardial infarction or one or more episodes of unstable angina within 6 months prior to enrollment
* Subjects with a history of malignant disease
* Subjects who are currently on chemotherapy treatment

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-01 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of the of device and/or procedure related adverse events
Evaluation of blood chemistry, hematology and urinalysis
Ability to record electrical activity from the stomach
Ability to communicate between patient wand and the device.

SECONDARY OUTCOMES:
Significant decrease in the HbA1c values between baseline and end-of-treatment
Reduction in the required medications due to improved glycemia.
Significant reduction in weight loss between baseline and end-of-treatment
Improvement in co-morbid parameters

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Ludvik, Prof., Principal Investigator — Allgemeinen Krankenhauses der Stadt Wein AkH
Locations (1):
- Allgemeinen Krankenhauses der Stadt Wein AkH, Vienna, Austria